CLINICAL TRIAL: NCT02749526
Title: Endostar Combined With MPFC Adjuvant Treatment of Esophageal Cancer Clinical Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual rate
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-ENDO-003
Record Dates: First submitted 2016-03-28; First posted 2016-04-25 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Esophageal
Keywords: Recombinant human endostatin，Endo
MeSH Terms: interventions — endostar protein; Cisplatin; gimeracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endostar combined with MPFC (Experimental): Chemotherapy regimens (er degree + mPFC) :
  Endostar:
  degrees 30 mg civ24h d0-6;
  Liposo:
  135 mg/m2 D1; cisplatin: D1-3, 25 mg/m2
  Gimeracil and Oteracil Potassium (Tegafur):
  (40 mg bid Tegafur), D1-14. A course of 3 weeks, after two course of chemotherapy the CT/MR/ultrasonic gastroscopy.
  Interventions: Drug: "Endostar"; Drug: Liposo; Drug: cisplatin; Drug: Gimeracil and Oteracil Potassium （Tegafur）

INTERVENTIONS:
Drug: "Endostar" — 30mg civ24h d0-6.A course of 3 weeks, after two course of chemotherapy the CT/MR/ultrasonic gastroscopy.
Drug: Liposo — 135mg/m2 D1.A course of 3 weeks, after two course of chemotherapy the CT/MR/ultrasonic gastroscopy.
Drug: cisplatin — 25mg/m2 D1-3.A course of 3 weeks, after two course of chemotherapy the CT/MR/ultrasonic gastroscopy.
Drug: Gimeracil and Oteracil Potassium （Tegafur） — 40mg bid，D1-14.A course of 3 weeks, after two course of chemotherapy the CT/MR/ultrasonic gastroscopy.

SUMMARY:
Endostar ® (recombinant human endostatin) continuous intravenous infusion combined with mPFC neoadjuvant treatment of esophageal cancer arm, Ⅱ single-center clinical trial.

DETAILED DESCRIPTION:
1. Research purpose: Endostar (recombinant human endostatin) continuous intravenous infusion combined with chemotherapy for stage Ⅲ resectable or potentially resectable esophageal cancer efficacy and safety and to maintain the efficacy and safety.
2. The main objectives: R0 resection rate

Secondary objectives:

1. pCR rate
2. 3-year disease-free survival
3. Security and complications
4. DFS, OS
5. Quality of Life

3.The number of research centers and research time: This study intends to preside and implemented by the Jiangsu Provincial People's Hospital, Professor Gu Yanhong. The trial is scheduled to start in September 2015, planned to stop in June 2016 into the group, one patient surgery follow-up to the last end, get the primary endpoint and safety, surgical complications secondary endpoint. This study will continue to follow-up the patient DFS, OS and other secondary end points.

ELIGIBILITY:
Inclusion Criteria:

* patients with esophageal cancer confirmed by histology or cytology;
* according to TNM staging for Ⅲ period, previous untreated can be removed and potentially resectable esophageal cancer patients;
* can eat more than liquid diet;No signs before esophageal perforation;No distant metastasis;
* male or female, age 18 and 75 years old or less or more;
* ECOG PS 0 ~ 1 minute;
* is expected to survive period for 3 months or more,
* enough blood function: absolute neutrophil count (ANC) or 2 x 109 / L and the • platelet count 100 x 109 / L or higher acuity 9 g/dL and hemoglobin;Liver function
* enough: upper limit of total bilirubin acuities were normal (ULN);AST and ALT acuities were 2.5 times the upper limit of normal (ULN);Alkaline phosphatase 5 times the upper limit of normal or less (ULN);
* enough renal function, serum creatinine or less normal limit (ULN) or calculated creatinine clearance or 60 mL/min.
* basic normal ecg, no healing trauma;
* always not received anti-tumor drug treatment;
* ever had had surgery patients, request to study treatment began to have more than 4 weeks, and the patient has recovered;
* a complete uterus of female in the group within 28 days before the study must have a negative pregnancy test results (except amenorrhea has 24 months).If the pregnancy test from the first time for more than 7 days, is the need for urine pregnancy test validation (within 7 days before the first delivery).
* prior to biological agents, especially e. coli genetically engineered products without severe allergic reactions;

Exclusion Criteria:

* there is a clear taxol allergy history;
* pregnancy, nursing mothers, or have fertility but not women using contraception;
* the existing serious acute infection, and not be controlled;Or fester sex and chronic infection, wound in delay no more;
* the original serious heart disease, including: higher risk of congestive heart failure, unable to control arrhythmia, unstable angina, myocardial infarction, severe valvular heart disease, and resistant hypertension;
* is not easy to control nerve, mental illness or mental disorders, compliance is poor, can't cooperate with accounts and response to treatment;Primary brain tumors or CNS metastases illness did not get a control, has obvious symptoms in cranial hypertension or nerve spirit;
* with bleeding tendency;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
R0 Resection rate | up to 8 months

SECONDARY OUTCOMES:
pCR rate | up to 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Gu Yanhong, PI, Study Chair — China:Jiangsu people's hospital
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No